CLINICAL TRIAL: NCT06077643
Title: Workshops and Exchange Groups for Laryngectomized Patients
Acronym: GELAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP230743
Record Dates: First submitted 2023-10-05; First posted 2023-10-11 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Laryngectomy; Status; Laryngeal Cancer
Keywords: Laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exchange group: Each patient will participate in a cycle of four sessions, over four months. Each will be carried out with five patients, in order to facilitate exchanges. The aim is to organize eight groups that will each complete a cycle. This will allow to include about forty patients in the study.
- Control group: Patients who don't want to participate in the exchange groups but agree to be included in the control group. They will have to complete the quality of life questionnaires four months apart.
  Estimation of 10 patients included.

SUMMARY:
This research is conducted with the aim of improving the quality of life of laryngectomized patients and their entourage. Worldwide, there are 185,000 new cases of laryngeal cancer per year. In Europe, between 2000 and 2007, the crude annual incidence rates of these cancers were 4.6/100,000 with a 5-year survival rate of 61%.

In France, about 30 to 35% of cancers of the upper aerodigestive tract are localized to the larynx, or about 43,000 cases per year. Most patients are men (89%) between 50 and 70 years old. One of the treatments for these cancers is to perform an excision of the larynx thus removing the entire tumor, it is the total laryngectomy. The trachea is thus permanently removed from the skin and the digestive tract becomes independent.

DETAILED DESCRIPTION:
In the ENT department of Bichat Hospital, there is an average of fourteen surgeries of this type per year, over the last three years. The direct consequences of total laryngectomy are multiple:

* loss of phonation (voice) and need to learn to speak again through speech therapy;
* Disappearance of oral-nasal breathing (and therefore loss of smell, or even taste);
* Disappearance of the capacity of the effort with closed glottis (used in the acts of daily life: defecation, sexual act in men, etc.);
* Impairment of body image and sometimes self-esteem.

For these reasons, it is essential to accompany patients post-operative to help them understand their body image and mitigate the direct and indirect consequences of this intervention. There are very few organizations to assist these patients in this life change.

To support laryngectomized patients, the study will test and validate the creation of self-help and support groups. The study will include laryngectomized patients who wish and can participate in these groups.

The sessions will take place as follows:

* 1st: presentation of each, answers to questions;
* 2nd: intervention of the association of the mutilated of the voice;
* 3rd: questions / answers with a resource patient (laryngectomized for 13 years in Bichat);
* 4th: grouping of all participants to assess patient satisfaction.

To assess the benefit of these meetings, a global quality of life questionnaire (WHOQOL-BREF) and an ENT-specific questionnaire (EORTC QLQH&n43) will be given to patients before the first session and retrieved beforehand. The patient will be able to participate in the sessions only if the questionnaires are submitted. The questionnaires are accompanied by a free text part, so that the person fills in the keys that the workshops have brought him. Patients who cannot participate in the exchange groups for geographical or personal reasons will constitute a control group. They will also complete the two questionnaires four months apart. The number of patients registered and the participation rate at each session will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Have had a total laryngectomy at Bichat Hospital or HEGP within the last four years
* Have completed all the specific care of the pathology that required the total laryngectomy
* Be able to travel to Bichat Hospital for all four sessions
* Be over 18 years of age
* Have received informed information about the conduct of the research.

Exclusion Criteria:

* WHO simplified autonomy scale greater than 2, i.e. from normal activity to ambulant and able to take care of themselves, but unable to provide work and bedridden for less than 50% of their time
* Patient who does not speak or understand French
* Lack of affiliation to a social security scheme or CMU
* Patient benefiting from legal protection measures (guardianship or curatorship)
* Patient who has communicated an objection to their inclusion, after informed information.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who has benefited from a total laryngectomy in the ENT department of Bichat Hospital or Georges Pompidou European Hospital, less than four years ago.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
Differences in quality of life scores before and after the program, between the program and non-program control groups. | 4 months
  The aim is to show a difference in patients' overall quality of life scores via the WHOQOL-BREF questionnaire, before and after the program.

SECONDARY OUTCOMES:
For overall quality of life using the WHOQOL-BREF questionnaire, comparison of the average patient scores, before and after exchange groups. | 4 months
  The aim is to show a difference in patients' overall quality of life scores via the WHOQOL-BREF questionnaire, before and after the program.
For ENT-specific quality of life using the EORTC QLQH&n43 questionnaire, comparison of the average patient scores, before and after exchange groups. | 4 months
  The aim is to show a difference in quality of life scores specific to ENT EORTC QLQH&n43, before and after the program.
Evaluation of the participation rate (number of patients present out of the number of patients enrolled), during each session via the OVET software. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Angèle Germon, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat - Claude Bernard Hospital, Paris, France